CLINICAL TRIAL: NCT00539149
Title: Amoxycillin Versus Placebo for Resolution of Otitis Media With Effusion and Prevention of Acute Otitis Media With Perforation in Aboriginal Infants: a Randomised Controlled Trial.
Brief Title: Long-term Antibiotics for Treatment and Prevention of Otitis Media in Aborignal Children
Acronym: COMIT1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COMIT1; NHMRC 954086
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2007-10

CONDITIONS: Otitis Media
Keywords: Acute otitis media; Otitis media with effusion; Tympanic membrane perforation
MeSH Terms: conditions — Otitis Media; Otitis Media with Effusion; Tympanic Membrane Perforation | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Amoxycillin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo equivalent to amoxycillin

INTERVENTIONS:
Drug: Amoxycillin — 50 mg/kg/day twice daily
  Arms: 1
Drug: Placebo equivalent to amoxycillin — 50 mg/kg/d twice daily
  Arms: 2

SUMMARY:
This clinical trial was conducted in a population where tympanic membrane perforation occurs in 60% infants in the first year of life. Nasopharyngeal colonisation (nasal contamination) with pathogenic bacteria occurs within weeks of life and predicts persistent middle ear infection throughout childhood. The trial aimed to assess whether twice daily antibiotics commencing at first detection of middle ear effusion would cure the infection and/or prevent disease progression, compared to placebo.

The study was conducted in three remote Aboriginal communities in the Northern Territory of Australia. The annual birth cohort was 45.

Aboriginal infants were seen as soon as possible after birth, and at 2 weekly intervals until middle ear effusion was detected by pneumatic otoscopy and tympanometry. Following consent, infants were randomised to either amoxycillin(50 mg/kg/d BD) or placebo equivalent for up to 24 weeks, or until normal middle ear status was detected at 2 consecutive monthly scheduled examinations. At monthly examinations the infant also had a general health check, parents were interviewed, child's medical record was reviewed, and nasopharyngeal swabs were collected.

ELIGIBILITY:
Inclusion Criteria:

* Australian Aboriginal
* Living in participating remote community
* Less than 12 months of age

Exclusion Criteria:

* Less than 32 weeks gestation
* Chronic condition requiring continuous antibiotic
* Ear, nose or throat abnormality

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 1996-04; Study Completion 2001-03 (Actual)

PRIMARY OUTCOMES:
Proportion of children with middle ear effusion | end of intervention
Proportion of study visits at which middle ear effusion detected | during intervention

SECONDARY OUTCOMES:
Proportion of infants with tympanic membrane perforation | end of intervention
Proportion of study visits with tympanic membrane perforation | during intervention
Proportion of infants with nasopharyngeal colonisation with resistant Streptococcus pneumoniae | end of intervention
proportion of infants withdrawn from study due to intervention adverse events | end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: John D Mathews, PhD, DSc., Principal Investigator — Menzies School of Health Research and University of Melbourne
Locations (1):
- Menzies School of Health Research, Darwin, Northern Territory, Australia

REFERENCES:
- [Background] Leach AJ, Morris PS. Antibiotics for the prevention of acute and chronic suppurative otitis media in children. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD004401. doi: 10.1002/14651858.CD004401.pub2. PMID 17054203
- [Background] Morris PS, Leach AJ, Halpin S, Mellon G, Gadil G, Wigger C, Mackenzie G, Wilson C, Gadil E, Torzillo P. An overview of acute otitis media in Australian Aboriginal children living in remote communities. Vaccine. 2007 Mar 22;25(13):2389-93. doi: 10.1016/j.vaccine.2006.09.006. Epub 2006 Sep 22. PMID 17030497
- [Background] Morris PS, Leach AJ, Silberberg P, Mellon G, Wilson C, Hamilton E, Beissbarth J. Otitis media in young Aboriginal children from remote communities in Northern and Central Australia: a cross-sectional survey. BMC Pediatr. 2005 Jul 20;5:27. doi: 10.1186/1471-2431-5-27. PMID 16033643
- [Background] Leach AJ, Morris PS. Perspectives on infective ear disease in indigenous Australian children. J Paediatr Child Health. 2001 Dec;37(6):529-30. doi: 10.1046/j.1440-1754.2001.00729.x. PMID 11903828
- [Background] Coates HL, Morris PS, Leach AJ, Couzos S. Otitis media in Aboriginal children: tackling a major health problem. Med J Aust. 2002 Aug 19;177(4):177-8. doi: 10.5694/j.1326-5377.2002.tb04727.x. No abstract available. PMID 12175319
- [Result] Leach AJ, Morris PS, Smith-Vaughan H, Mathews JD. In vivo penicillin MIC drift to extremely high resistance in Serotype 14 Streptococcus pneumoniae persistently colonizing the nasopharynx of an infant with chronic suppurative lung disease: a case study. Antimicrob Agents Chemother. 2002 Nov;46(11):3648-9. doi: 10.1128/AAC.46.11.3648-3649.2002. PMID 12384383
- [Derived] Mulvaney CA, Galbraith K, Webster KE, Rana M, Connolly R, Marom T, Daniel M, Venekamp RP, Schilder AG, MacKeith S. Antibiotics for otitis media with effusion (OME) in children. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD015254. doi: 10.1002/14651858.CD015254.pub2. PMID 37870130